CLINICAL TRIAL: NCT00463138
Title: Follow-up Study on Recipients of Treatment at the Jerusalem Center for the Treatment of Psychotrauma
Status: Completed | Type: Observational
Sponsor: Herzog Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ruth Pat-Horenzcyk, Research director, Herzog Hospital
Other Study IDs: Brom3CTIL
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: perceived increase or decrease in symptoms post treatment; Satisfaction with the treatment
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Crisis intervention

SUMMARY:
Researchers examined perceived satisfaction and perceived increase or decrease in symptoms among recipients of treatment at the Jerusalem Center for the Treatment of Psychotrauma, using self report methods. Researchers hypothesized that a significant number of recipients would report a decrease in their symptoms and general satisfaction with the treatment they received.

DETAILED DESCRIPTION:
Researchers conducted a follow-up study of clients of Meytiv, the clinical branch of the Jerusalem Center for the Treatment of Psychotrauma. Researchers plan to use the results of the study to better understand the demographics of those who come to the Center, and to improve the services offered to our clients. Before beginning treatment, every Meytiv client filled out a questionnaire in which information is requested regarding demographics, trauma history, symptoms, and various levels of functioning. Researchers administered a similar self-report questionnaire to all clients upon completion of treatment. The follow-up questionnaire contained the following several indices: the Traumatic Events Screening Inventory (TESI), which requests a client's trauma history; the Multidimensional Scale of Perceived Social Support, which measures level of family, friend, and other support; the Brief Symptom Inventory, which measures level of various psychiatric symptoms, including somatic complaints, depressive symptoms, anxiety, and paranoid or hostile thoughts; the Self-Efficacy Scale, which measures level of self-reliance and confidence in one's ability to cope with stressors; and PDS, which measures subjective response to trauma, symptoms, and and level of functioning. This questionnaire, which mirrors one completed by all Meytiv's clients before treatment, was administered to those clients who completed treatment within a year of the study. Clients completed the follow-up questionnaire on condition that if they were in need of further treatment, Meytiv would refer them to the appropriate provider. Responses will be coded and analyzed to check significance among potentially related variables, including demographic variables. Most importantly, results of the follow-up questionnaire will be compared to its parallel from the beginning of treatment in order to examine what effects our treatment has on one's symptoms, and whether our clients have been satisfied

ELIGIBILITY:
Inclusion Criteria:

* All clients who were exposed to a traumatic event within the last 2 years and completed treatment at the Trauma Center within the last year

Exclusion Criteria:

* Clients under the age of 12

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All clients who were exposed to a traumatic event within the last 2 years and completed treatment at the Trauma Center within the last year
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
depressive symptoms, anxiety, PDS, which measures subjective response to trauma, symptoms, and and level of functioning. | April 2007- March 2008

SECONDARY OUTCOMES:
level of family, friend, and other support, Self-Efficacy Scale | Aprol 2007- March2008

OTHER OUTCOMES:
Traumatic Events Screening Inventory (TESI) | April 2008- March 2008

CONTACTS AND LOCATIONS:
Overall Officials: Danny Brom, Ph.D, Principal Investigator — Israel Center for the Treatment of Psychotrauma